CLINICAL TRIAL: NCT00661661
Title: A Long-term, Open-label Study Of Cp-690,550 to Confirm The Safety Following Long Term Administration Of Cp-690,550 In The Treatment Of Rheumatoid Arthritis
Brief Title: Long-Term, Open-Label Study Of CP-690,550 For Treatment Of Rheumatoid Arthritis In Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3921041
Record Dates: First submitted 2008-02-07; First posted 2008-04-18 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Long term open label study in Japan; CP-690; 550; tofacitinib
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CP-690,550 (Experimental)
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — 5 mg BID up to 10 mg BID until launch

SUMMARY:
The purpose of this study is to determine the long-term effectiveness and safety of CP-690,550 for the treatment of rheumatoid arthritis. Subjects are only eligible for this study after they have completed participation in another "qualifying" study of CP-690,550.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed their participation in a randomized "qualifying" study of CP-690,550 for the treatment of rheumatoid arthritis

Exclusion Criteria:

* Serious medical conditions that would make treatment with CP-690,550 potentially unsafe

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2008-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (56):
- Japan (56):
  - National hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Chiba-East Hospital, Chiba, Chiba
  - Chiba-ken Saiseikai Narashino Hospital, Narashino, Chiba
  - Shimoshizu National Hospital, Yotukaidou, Chiba
  - Kondo clinic for rheumatism and orthopaedics, Fukuoka, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Medical Co.LTA PS Clinic, Fukuoka, Fukuoka
  - Aso Iizuka Hospital, Iiduka, Fukuoka
  - University of Occupational and Environmental Health Hospital, Kitakyushu, Fukuoka
  - St. Mary's Hospital, Kurume, Fukuoka
  - SHONO Rheumatism Clinic, Sawara-ku, Fukuoka
  - Fukusima Daiichi Hospital, Fukushima, Fukushima
  - Inoue Hospital, Takasaki, Gunma
  - Higashihiroshima Memorial Hospital, Higashihiroshima, Hiroshima
  - Hiroshima Rheumatology Clinic, Hiroshima, Hiroshima
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima, Hiroshima
  - Katayama Orthopedic Rheumatology Clinic, Asahikawa, Hokkaido
  - Sapporo city general hospital, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hokkaido Medical Center for Rheumatic Diseases, Sapporo, Hokkaido
  - The Hospital of Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Taga General Hospital, Hitachi-shi, Ibaraki
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - Keio University Hospital, Shinjuku-ku, Tokyo, Japan
  - National Hospital Organization Sagamihara National Hospital, Sagamihara, Kanagawa
  - Kumamoto Saishunso National Hospital, Koushi, Kumamoto
  - Kumamoto Orthopaedic Hospital, Kumamoto, Kumamoto
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - National hospital Organization Mie Chuou Medical Center, Tsu, Mie-ken
  - Hikarigaoka Spellman Hospital, Sendai, Miyagi
  - Nagasaki University Hospital of Medicine and Dentistry, Nagasaki, Nagasaki
  - National Hospital Organization Nagasaki Medical Center, Ohmura, Nagasaki
  - Sasebo Chuo Hospital, Sasebo, Nagasaki
  - Higami hospital, Kashihara, Nara
  - Niigata University Medical & Dental Hospital, Niigata, Niigata
  - A Medical Corporation Oribe Rheumatism Internist Clinic, Ōita, Oita Prefecture
  - National Hospital Organization Osaka Minami Center, Kawachi-Nagano, Osaka
  - The Tazuke Kofukai Medical Research Institute Kitano Hospital, Osaka, Osaka
  - Ureshino Medical Center, Ureshino, Saga-ken
  - Saitama Medical Center, Kawagoe-shi, Saitama
  - Kitasato University Kitasato Institute Medical Center Hospital, Kitamoto, Saitama
  - Saitama city hospital, Saitama, Saitama
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Tokyo Women's Medical University Medical Center East, Arakawa-ku, Tokyo
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Medical And Dental University Hospital, Faculty of Medicine, Bunkyo-ku, Tokyo
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - Sasaki Foundation Kyoundo Hospital, Chiyoda-ku, Tokyo
  - Juntendo Tokyo Koto Geriatric Medical Center, Koto-ku, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - National Hospital Organization MURAYAMA Medical Center, Musashimurayama-shi, Tokyo
  - Fukuhara Hospital, Setagaya-ku, Tokyo
  - Tokyo Women's Medical University, Institute of Rheumatology, Shinjyuku-ku, Tokyo
  - Sendai Taihaku Hospital, Miyagi

REFERENCES:
- [Derived] Strand V, Schulze-Koops H, Al-Emadi S, Kinch CD, Gruben D, Germino R, Connell CA, Mysler E. Sex differences in the efficacy, safety and persistence of tofacitinib in patients with rheumatoid arthritis: a post hoc analysis of phase III and long-term extension trials. BMJ Open. 2025 Dec 24;15(12):e082366. doi: 10.1136/bmjopen-2023-082366. PMID 41448717
- [Derived] Pope J, Finckh A, Silva-Fernandez L, Mandl P, Fan H, Rivas JL, Valderrama M, Montoro M. Tofacitinib Monotherapy in Rheumatoid Arthritis: Clinical Trials and Real-World Data Contextualization of Patients, Efficacy, and Treatment Retention. Open Access Rheumatol. 2024 Jun 11;16:115-126. doi: 10.2147/OARRR.S446431. eCollection 2024. PMID 38883150
- [Derived] Curtis JR, Wollenhaupt J, Tas SW, Chatzidionysiou K, Wang L, Roberts K, Tsekouras V. Determinants of tofacitinib discontinuation in adult patients with rheumatoid arthritis during long-term extension studies up to 9.5 years. Rheumatol Adv Pract. 2024 May 11;8(2):rkae063. doi: 10.1093/rap/rkae063. eCollection 2024. PMID 38854417
- [Derived] Charles-Schoeman C, Hyde C, Guan S, Parikh N, Wang J, Shahbazian A, Stockert L, Andrews J. Relationship Between Paraoxonase-1 Genotype and Activity, and Major Adverse Cardiovascular Events and Malignancies in Patients With Rheumatoid Arthritis Receiving Tofacitinib. J Rheumatol. 2023 Jul 15:jrheum.2023-0112. doi: 10.3899/jrheum.2023-0112. Online ahead of print. PMID 37453736
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] van der Heijde D, Landewe RBM, Wollenhaupt J, Strengholt S, Terry K, Kwok K, Wang L, Cohen S. Assessment of radiographic progression in patients with rheumatoid arthritis treated with tofacitinib in long-term studies. Rheumatology (Oxford). 2021 Apr 6;60(4):1708-1716. doi: 10.1093/rheumatology/keaa476. PMID 33057725
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Fleischmann R, Wollenhaupt J, Takiya L, Maniccia A, Kwok K, Wang L, van Vollenhoven RF. Safety and maintenance of response for tofacitinib monotherapy and combination therapy in rheumatoid arthritis: an analysis of pooled data from open-label long-term extension studies. RMD Open. 2017 Dec 18;3(2):e000491. doi: 10.1136/rmdopen-2017-000491. eCollection 2017. PMID 29435359
- [Derived] Fleischmann R, Wollenhaupt J, Cohen S, Wang L, Fan H, Bandi V, Andrews J, Takiya L, Bananis E, Weinblatt ME. Effect of Discontinuation or Initiation of Methotrexate or Glucocorticoids on Tofacitinib Efficacy in Patients with Rheumatoid Arthritis: A Post Hoc Analysis. Rheumatol Ther. 2018 Jun;5(1):203-214. doi: 10.1007/s40744-018-0093-7. Epub 2018 Feb 7. PMID 29417430
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Yamanaka H, Tanaka Y, Takeuchi T, Sugiyama N, Yuasa H, Toyoizumi S, Morishima Y, Hirose T, Zwillich S. Tofacitinib, an oral Janus kinase inhibitor, as monotherapy or with background methotrexate, in Japanese patients with rheumatoid arthritis: an open-label, long-term extension study. Arthritis Res Ther. 2016 Jan 28;18:34. doi: 10.1186/s13075-016-0932-2. PMID 26818974
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921041&StudyName=Long-Term%2C%20Open-Label%20Study%20Of%20CP-690%2C550%20For%20Treatment%20Of%20Rheumatoid%20Arthritis%20In%20Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received study drug (CP-690,550 or placebo) in the precedent study A3921039 (NCT00603512) for 12 weeks, A3921040 (NCT00687193) for 12 weeks, or A3921044 (NCT00847613) for 2 years.
Groups:
- CP-690,550 5 mg BID: CP-690,550 5 milligram (mg) tablet orally twice daily (BID). After Week 12, the dose could be changed 5 mg BID or 10 mg BID based on investigator discretion. This study was continued until CP-690,550 was commercially supplied to participants at the sites. Participants who were exposed to 10 mg BID for less than 84 days in total within the current study (A3921041) were grouped into CP-690,550 5 mg BID.
- CP-690,550 10 mg BID: CP-690,550 5 milligram (mg) tablet orally twice daily (BID). After Week 12, the dose could be changed 5 mg BID or 10 mg BID based on investigator discretion. This study was continued until CP-690,550 was commercially supplied to participants at the sites. Participants who were exposed to 10 mg BID for more than or equal to 84 days in total within the long-term safety study (A3921041) were grouped into CP-690,550 10 mg BID.
Period: Overall Study
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID
Started | 382 | 105
Completed | 242 | 66
Not Completed | 140 | 39
Not completed — Adverse Event | 99 | 24
Not completed — Lack of Efficacy | 3 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 15 | 5
Not completed — Other | 22 | 7
Not completed — Not assigned treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (11.2) | 49.3 (11.7) | 52.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 318 | 86 | 404
  Male | 63 | 19 | 82

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response
Description: ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in tender joint count; >=20% improvement in swollen joint count; and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP). The baseline data of Study A3921039, A3921040 or A3921044 were used as baseline data for efficacy evaluations except for Modified Total Sharp Score (mTSS).
Time Frame: Weeks 2, 4,8,12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276 and 288
Population: Full analysis set (FAS): All participants who received at least 1 dose of study medication in current study. No imputation was used (observed data).
Measure: Number; unit: Percentage of participants
Groups:
- Total: All subjects were assigned oral CP-690,550 5 mg tablets twice a day at baseline visit. Dose flexibility (increasing from 5 mg BID to 10 mg BID, reducing from 10 mg BID to 5 mg BID, or temporary discontinuation) during study was allowed in consideration for the risks and benefits to the patient's condition. Data was summarized in three reporting groups including CP-690,550 5 mg BID, CP-690,550 10 mg BID and Total.
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Percentage of participants
  Week 2 (n= 378, 105, 483) | 80.2 | 68.6 | 77.6
  Week 4 (n=373, 105, 478) | 87.1 | 70.5 | 83.5
  Week 8 (n=371, 105, 476) | 90.0 | 72.4 | 86.1
  Week 12 (n=370, 105, 475) | 91.9 | 77.1 | 88.6
  Week 24 (n=357, 104, 461) | 90.8 | 85.6 | 89.6
  Week 36 (n=339, 102, 441) | 94.1 | 87.3 | 92.5
  Week 48 (n=331, 102, 433) | 93.7 | 88.2 | 92.4
  Week 60 (n=323, 102, 425) | 92.3 | 90.2 | 91.8
  Week 72 (n=315, 99, 414) | 92.4 | 86.9 | 91.1
  Week 84 (n=309, 92, 401) | 93.2 | 87.0 | 91.8
  Week 96 (n=281, 87, 368) | 92.2 | 92.0 | 92.1
  Week 108 (n=259, 84, 343) | 91.9 | 86.9 | 90.7
  Week 120 (n=242, 80, 322) | 91.3 | 88.8 | 90.7
  Week 132 (n=232, 79, 311) | 92.2 | 84.8 | 90.4
  Week 144 (n=224, 76, 300) | 89.7 | 86.8 | 89.0
  Week 156 (n=219, 73, 292) | 91.3 | 84.9 | 89.7
  Week 168 (n=213, 70, 283) | 92.5 | 82.9 | 90.1
  Week 180 (n=180, 57, 237) | 92.8 | 86.0 | 91.1
  Week 192 (n=138, 42, 180) | 92.8 | 85.7 | 91.1
  Week 204 (n=109, 30, 139) | 92.7 | 90.0 | 92.1
  Week 216 (n=76, 13, 89) | 96.1 | 84.6 | 94.4
  Week 228 (n=68, 5, 73) | 91.2 | 80.0 | 90.4
  Week 240 (n=65, 5, 70) | 93.8 | 80.0 | 92.9
  Week 252 (n=65, 5, 70) | 92.3 | 80.0 | 91.4
  Week 264 (n=59, 5, 64) | 89.8 | 80.0 | 89.1
  Week 276 (n=22, 1, 23) | 95.5 | 100 | 95.7
  Week 288 (n=3, 0, 3) | 100 | 0 | 100

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: ACR50 response: greater than or equal to (>=) 50 percent (%) improvement in tender joint count; >=50% improvement in swollen joint count; and >=50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP). The baseline data of Study A3921039, A3921040 or A3921044 were used as baseline data for efficacy evaluations except for Modified Total Sharp Score (mTSS).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Percentage of participants
  Week 2 (n= 378, 105, 483) | 59.5 | 36.2 | 54.5
  Week 4 (n=373, 105, 478) | 63.8 | 35.2 | 57.5
  Week 8 (n=371, 105, 476) | 70.4 | 47.6 | 65.3
  Week 12 (n=370, 105, 475) | 70.8 | 46.7 | 65.5
  Week 24 (n=357, 104, 461) | 76.2 | 62.5 | 73.1
  Week 36 (n=339, 102, 441) | 77.3 | 56.9 | 72.6
  Week 48 (n=331, 102, 433) | 77.3 | 59.8 | 73.2
  Week 60 (n=323, 102, 425) | 77.1 | 66.7 | 74.6
  Week 72 (n=315, 99, 414) | 77.8 | 74.7 | 77.1
  Week 84 (n=309, 92, 401) | 78.6 | 64.1 | 75.3
  Week 96 (n=281, 87, 368) | 78.3 | 60.9 | 74.2
  Week 108 (n=259, 84, 343) | 79.9 | 72.6 | 78.1
  Week 120 (n=242, 80, 322) | 76.4 | 68.8 | 74.5
  Week 132 (n=232, 79, 311) | 77.2 | 72.2 | 75.9
  Week 144 (n=224, 76, 300) | 78.1 | 69.7 | 76.0
  Week 156 (n=219, 73, 292) | 79.5 | 65.8 | 76.0
  Week 168 (n=213, 70, 283) | 79.3 | 67.1 | 76.3
  Week 180 (n=180, 57, 237) | 82.2 | 71.9 | 79.7
  Week 192 (n=138, 42, 180) | 79.7 | 61.9 | 75.6
  Week 204 (n=109, 30, 139) | 84.4 | 80.0 | 83.5
  Week 216 (n=76, 13, 89) | 86.8 | 53.8 | 82.0
  Week 228 (n=68, 5, 73) | 76.5 | 80.0 | 76.7
  Week 240 (n=65, 5, 70) | 83.1 | 40.0 | 80.0
  Week 252 (n=65, 5, 70) | 86.2 | 40.0 | 82.9
  Week 264 (n=59, 5, 64) | 84.7 | 40.0 | 81.3
  Week 276 (n=22, 1, 23) | 81.8 | 100 | 82.6
  Week 288 (n=3, 0, 3) | 100 | 0 | 100

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response: greater than or equal to (>=) 70 percent (%) improvement in tender joint count; >=70% improvement in swollen joint count; and >=70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP). The baseline data of Study A3921039, A3921040 or A3921044 were used as baseline data for efficacy evaluations except for Modified Total Sharp Score (mTSS).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Percentage of participants
  Week 2 (n= 378, 105, 483) | 37.0 | 19.0 | 33.1
  Week 4 (n=373, 105, 478) | 44.8 | 20.2 | 39.3
  Week 8 (n=371, 105, 476) | 47.7 | 21.0 | 41.8
  Week 12 (n=370, 105, 475) | 50.0 | 16.2 | 42.5
  Week 24 (n=357, 104, 461) | 54.1 | 27.9 | 48.2
  Week 36 (n=339, 102, 441) | 56.6 | 24.5 | 49.2
  Week 48 (n=331, 102, 433) | 59.8 | 34.3 | 53.8
  Week 60 (n=323, 102, 425) | 59.1 | 37.3 | 53.9
  Week 72 (n=315, 99, 414) | 61.9 | 38.4 | 56.3
  Week 84 (n=309, 92, 401) | 60.2 | 35.9 | 54.6
  Week 96 (n=281, 87, 368) | 59.4 | 42.5 | 55.4
  Week 108 (n=259, 84, 343) | 60.6 | 42.9 | 56.3
  Week 120 (n=242, 80, 322) | 62.0 | 37.5 | 55.9
  Week 132 (n=232, 79, 311) | 60.8 | 40.5 | 55.6
  Week 144 (n=224, 76, 300) | 61.2 | 35.5 | 54.7
  Week 156 (n=219, 73, 292) | 61.6 | 41.1 | 56.5
  Week 168 (n=213, 70, 283) | 62.9 | 41.4 | 57.6
  Week 180 (n=180, 57, 237) | 63.9 | 47.4 | 59.9
  Week 192 (n=138, 42, 180) | 63.8 | 42.9 | 58.9
  Week 204 (n=109, 30, 139) | 62.4 | 56.7 | 61.2
  Week 216 (n=76, 13, 89) | 69.7 | 30.8 | 64.0
  Week 228 (n=68, 5, 73) | 63.2 | 20.0 | 60.3
  Week 240 (n=65, 5, 70) | 69.2 | 20.0 | 65.7
  Week 252 (n=65, 5, 70) | 73.8 | 20.0 | 70.0
  Week 264 (n=59, 5, 64) | 71.2 | 20.0 | 67.2
  Week 276 (n=22, 1, 23) | 68.2 | 0 | 65.2
  Week 288 (n=3, 0, 3) | 66.7 | 0 | 66.7

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom, arise, eat, walk, reach, grip, hygiene and common activities over past week. Each item scored on 4-point scale, 0 to 3: 0=no difficulty; 1=some difficulty;2=much difficulty; 3=unable to do. Overall score was computed as sum of domain sc ores and divided by number of domains answered. Total possible score range 0-3: 0=least difficulty and 3=extreme difficulty. The baseline data of Study A3921039, A3921040 or A3921044 were used as baseline data for efficacy evaluations except for Modified Total Sharp Score (mTSS).
Time Frame: Baseline, Weeks 2, 4,8,12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276 and 288
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 2 (n= 378, 105, 483) | -0.55 (0.03) | -0.44 (0.05) | -0.53 (0.03)
  Week 4 (n=372, 105, 477) | -0.61 (0.03) | -0.45 (0.05) | -0.57 (0.03)
  Week 8 (n=371, 105, 476) | -0.66 (0.03) | -0.49 (0.05) | -0.62 (0.03)
  Week 12 (n=370, 105, 475) | -0.66 (0.03) | -0.51 (0.05) | -0.63 (0.03)
  Week 24 (n=357, 104, 461) | -0.69 (0.03) | -0.55 (0.05) | -0.65 (0.03)
  Week 36 (n=339, 102, 441) | -0.70 (0.03) | -0.54 (0.05) | -0.66 (0.03)
  Week 48 (n=331, 102, 433) | -0.70 (0.03) | -0.62 (0.05) | -0.68 (0.03)
  Week 60 (n=323, 102, 425) | -0.71 (0.03) | -0.57 (0.05) | -0.67 (0.03)
  Week 72 (n=315, 99, 414) | -0.72 (0.03) | -0.60 (0.05) | -0.69 (0.03)
  Week 84 (n=309, 92, 401) | -0.72 (0.04) | -0.61 (0.05) | -0.69 (0.03)
  Week 96 (n=281, 87, 368) | -0.72 (0.04) | -0.61 (0.06) | -0.69 (0.03)
  Week 108 (n=259, 84, 343) | -0.70 (0.04) | -0.64 (0.06) | -0.69 (0.03)
  Week 120 (n=242, 80, 322) | -0.70 (0.04) | -0.63 (0.06) | -0.68 (0.03)
  Week 132 (n=232, 79, 311) | -0.70 (0.04) | -0.64 (0.06) | -0.68 (0.03)
  Week 144 (n=224, 76, 300) | -0.67 (0.04) | -0.59 (0.07) | -0.65 (0.04)
  Week 156 (n=219, 72, 291) | -0.68 (0.04) | -0.62 (0.06) | -0.66 (0.03)
  Week 168 (n=213, 70, 283) | -0.68 (0.04) | -0.57 (0.07) | -0.65 (0.04)
  Week 180 (n=180, 57, 237) | -0.70 (0.05) | -0.63 (0.08) | -0.68 (0.04)
  Week 192 (n=138, 42, 180) | -0.69 (0.05) | -0.61 (0.09) | -0.67 (0.05)
  Week 204 (n=109, 30, 139) | -0.67 (0.06) | -0.67 (0.09) | -0.67 (0.05)
  Week 216 (n=76, 13, 89) | -0.62 (0.06) | -0.42 (0.09) | -0.59 (0.05)
  Week 228 (n=68, 5, 73) | -0.62 (0.06) | -0.25 (0.10) | -0.59 (0.06)
  Week 240 (n=65, 5, 70) | -0.66 (0.06) | -0.33 (0.14) | -0.64 (0.06)
  Week 252 (n=65, 5, 70) | -0.68 (0.07) | -0.25 (0.12) | -0.65 (0.06)
  Week 264 (n=59, 5, 64) | -0.65 (0.07) | -0.23 (0.07) | -0.62 (0.07)
  Week 276 (n=22, 1, 23) | -0.83 (0.11) | -0.63 (NA) — Standard error was not calculated due to one participant data available. | -0.82 (0.11)
  Week 288 (n=3, 0, 3) | -0.96 (0.37) | NA (NA) — Mean and standard error were not calculated because no data were available. | -0.96 (0.37)

5. Secondary Outcome: Change From Baseline in Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR])
Description: DAS28-4 (ESR) calculated from swollen joint count (SJC) and tender/painful joint count (TJC) using 28 joint count, erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PtGA) of disease activity (transformed score ranging 0 to 10; higher score indicated greater affectation due to disease activity). Total score range:0 to 9.4, higher score indicated more disease activity. The baseline data of Study A3921039, A3921040 or A3921044 were used as baseline data for efficacy evaluations except for Modified Total Sharp Score (mTSS).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 2 (n= 378, 105, 483) | -2.60 (0.07) | -1.94 (0.13) | -2.45 (0.06)
  Week 4 (n=372, 105, 477) | -2.77 (0.07) | -1.95 (0.13) | -2.59 (0.06)
  Week 8 (n=371, 104, 475) | -2.95 (0.06) | -2.14 (0.12) | -2.77 (0.06)
  Week 12 (n=370, 105, 475) | -3.01 (0.06) | -2.08 (0.12) | -2.81 (0.06)
  Week 24 (n=357, 104, 461) | -3.12 (0.06) | -2.42 (0.12) | -2.96 (0.06)
  Week 36 (n=339, 102, 441) | -3.18 (0.07) | -2.54 (0.13) | -3.03 (0.06)
  Week 48 (n=331, 102, 433) | -3.20 (0.07) | -2.72 (0.13) | -3.08 (0.06)
  Week 60 (n=323, 101, 424) | -3.25 (0.07) | -2.80 (0.12) | -3.15 (0.06)
  Week 72 (n=315, 99, 414) | -3.20 (0.07) | -2.83 (0.12) | -3.11 (0.06)
  Week 84 (n=309, 92, 401) | -3.26 (0.07) | -2.86 (0.14) | -3.17 (0.06)
  Week 96 (n=281, 87, 368) | -3.21 (0.07) | -2.87 (0.14) | -3.13 (0.07)
  Week 108 (n=259, 83, 342) | -3.22 (0.08) | -2.83 (0.15) | -3.12 (0.07)
  Week 120 (n=242, 79, 321) | -3.24 (0.08) | -2.78 (0.14) | -3.12 (0.07)
  Week 132 (n=232, 79, 311) | -3.14 (0.08) | -2.84 (0.15) | -3.07 (0.07)
  Week 144 (n=224, 76, 300) | -3.17 (0.09) | -2.84 (0.16) | -3.09 (0.08)
  Week 156 (n=218, 72, 290) | -3.08 (0.09) | -2.84 (0.16) | -3.02 (0.08)
  Week 168 (n=213, 70, 283) | -3.16 (0.09) | -2.87 (0.17) | -3.09 (0.08)
  Week 180 (n=178, 56, 234) | -3.21 (0.10) | -3.06 (0.19) | -3.18 (0.09)
  Week 192 (n=138, 42, 180) | -3.17 (0.11) | -3.07 (0.19) | -3.15 (0.09)
  Week 204 (n=109, 30, 139) | -3.24 (0.12) | -3.35 (0.25) | -3.26 (0.11)
  Week 216 (n=76, 13, 89) | -3.20 (0.13) | -2.44 (0.44) | -3.09 (0.13)
  Week 228 (n=68, 5, 73) | -3.08 (0.17) | -2.25 (0.58) | -3.02 (0.16)
  Week 240 (n=65, 5, 70) | -3.22 (0.15) | -2.61 (0.70) | -3.17 (0.14)
  Week 252 (n=65, 5, 70) | -3.33 (0.15) | -1.81 (0.51) | -3.23 (0.15)
  Week 264 (n=59, 5, 64) | -3.32 (0.15) | -2.09 (0.45) | -3.23 (0.14)
  Week 276 (n=21, 1, 22) | -3.34 (0.25) | -2.15 (NA) — Standard error was not calculated due to one participant data available. | -3.29 (0.24)
  Week 288 (n=3, 0, 3) | -2.95 (0.51) | NA (NA) — Mean and standard error were not calculated because no data were available. | -2.95 (0.51)

6. Secondary Outcome: Change From Baseline in Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP])
Description: DAS28-3 (CRP) was calculated from SJC and TJC using 28 joint count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. The baseline data of Study A3921039, A3921040 or A3921044 were used as baseline data for efficacy evaluations except for Modified Total Sharp Score (mTSS).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 2 (n= 378, 105, 483) | -2.44 (0.06) | -1.90 (0.12) | -2.32 (0.06)
  Week 4 (n=372, 105, 477) | -2.55 (0.06) | -1.90 (0.12) | -2.41 (0.06)
  Week 8 (n=371, 105, 476) | -2.68 (0.06) | -2.06 (0.11) | -2.55 (0.05)
  Week 12 (n=370, 105, 475) | -2.75 (0.06) | -1.97 (0.11) | -2.57 (0.05)
  Week 24 (n=357, 104, 461) | -2.85 (0.06) | -2.29 (0.11) | -2.72 (0.05)
  Week 36 (n=337, 102, 439) | -2.92 (0.06) | -2.45 (0.11) | -2.81 (0.05)
  Week 48 (n=331, 102, 433) | -2.92 (0.06) | -2.58 (0.12) | -2.84 (0.05)
  Week 60 (n=322, 102, 424) | -2.92 (0.06) | -2.60 (0.11) | -2.85 (0.05)
  Week 72 (n=315, 99, 414) | -2.93 (0.06) | -2.61 (0.11) | -2.86 (0.05)
  Week 84 (n=309, 92, 401) | -2.98 (0.06) | -2.70 (0.12) | -2.92 (0.06)
  Week 96 (n=281, 87, 368) | -2.95 (0.07) | -2.69 (0.13) | -2.88 (0.06)
  Week 108 (n=259, 83, 342) | -2.93 (0.07) | -2.64 (0.13) | -2.86 (0.06)
  Week 120 (n=242, 80, 322) | -2.97 (0.07) | -2.60 (0.13) | -2.88 (0.06)
  Week 132 (n=231, 79, 310) | -2.89 (0.07) | -2.66 (0.13) | -2.83 (0.06)
  Week 144 (n=224, 76, 300) | -2.90 (0.08) | -2.68 (0.14) | -2.85 (0.07)
  Week 156 (n=219, 72, 291) | -2.84 (0.08) | -2.70 (0.14) | -2.81 (0.07)
  Week 168 (n=213, 70, 283) | -2.90 (0.08) | -2.68 (0.15) | -2.84 (0.07)
  Week 180 (n=180, 57, 237) | -2.92 (0.09) | -2.80 (0.17) | -2.89 (0.08)
  Week 192 (n=138, 42, 180) | -2.93 (0.09) | -2.84 (0.16) | -2.91 (0.08)
  Week 204 (n=109, 30, 139) | -2.95 (0.11) | -3.05 (0.22) | -2.97 (0.10)
  Week 216 (n=76, 13, 89) | -2.94 (0.12) | -2.46 (0.34) | -2.87 (0.12)
  Week 228 (n=68, 5, 73) | -2.84 (0.17) | -2.38 (0.44) | -2.81 (0.16)
  Week 240 (n=65, 5, 70) | -2.97 (0.13) | -2.36 (0.57) | -2.92 (0.13)
  Week 252 (n=65, 5, 70) | -3.09 (0.14) | -1.89 (0.42) | -3.00 (0.14)
  Week 264 (n=58, 5, 63) | -3.13 (0.15) | -1.86 (0.30) | -3.03 (0.14)
  Week 276 (n=22, 1, 23) | -3.24 (0.24) | -1.50 (NA) — Standard error was not calculated due to one participant data available. | -3.16 (0.24)
  Week 288 (n=3, 0, 3) | -2.67 (0.27) | NA (NA) — Mean and standard error were not calculated because no data were available. | -2.67 (0.27)

7. Secondary Outcome: Change From Baseline in Patient Global Assessment of Arthritis
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm VAS where 0 = very well and 100 = very poorly. The baseline data of Study A3921039, A3921040 or A3921044 were used as baseline data for efficacy evaluations except for Modified Total Sharp Score (mTSS).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 2 (n= 378, 105, 483) | -34.52 (1.38) | -25.38 (2.43) | -32.54 (1.21)
  Week 4 (n=372, 105, 477) | -37.81 (1.36) | -25.34 (2.61) | -35.06 (1.23)
  Week 8 (n=371, 105, 476) | -39.61 (1.35) | -28.86 (2.31) | -37.24 (1.19)
  Week 12 (n=370, 105, 475) | -39.31 (1.38) | -27.33 (2.23) | -36.67 (1.20)
  Week 24 (n=357, 104, 461) | -40.67 (1.39) | -30.75 (2.53) | -38.43 (1.24)
  Week 36 (n=339, 102, 441) | -41.70 (1.42) | -29.95 (2.63) | -38.98 (1.27)
  Week 48 (n=331, 102, 433) | -41.03 (1.46) | -32.48 (2.56) | -39.02 (1.28)
  Week 60 (n=323, 102, 425) | -41.79 (1.44) | -34.33 (2.42) | -40.00 (1.25)
  Week 72 (n=315, 99, 414) | -41.30 (1.53) | -35.38 (2.31) | -39.88 (1.29)
  Week 84 (n=309, 92, 401) | -42.29 (1.53) | -35.12 (2.63) | -40.65 (1.33)
  Week 96 (n=281, 87, 368) | -41.90 (1.62) | -34.98 (2.88) | -40.27 (1.42)
  Week 108 (n=259, 84, 343) | -42.47 (1.67) | -34.95 (2.98) | -40.63 (1.46)
  Week 120 (n=242, 80, 322) | -42.97 (1.71) | -35.00 (3.05) | -40.99 (1.50)
  Week 132 (n=232, 79, 311) | -42.87 (1.73) | -35.05 (3.13) | -40.88 (1.52)
  Week 144 (n=224, 76, 300) | -42.48 (1.77) | -33.78 (3.22) | -40.27 (1.57)
  Week 156 (n=219, 72, 291) | -42.72 (1.71) | -32.64 (3.13) | -40.22 (1.52)
  Week 168 (n=213, 70, 283) | -43.00 (1.72) | -33.61 (3.22) | -40.67 (1.53)
  Week 180 (n=180, 57, 237) | -43.22 (1.91) | -36.14 (3.72) | -41.52 (1.71)
  Week 192 (n=138, 42, 180) | -42.05 (2.10) | -34.40 (3.95) | -40.27 (1.86)
  Week 204 (n=109, 30, 139) | -42.44 (2.36) | -35.73 (5.31) | -40.99 (2.18)
  Week 216 (n=76, 13, 89) | -42.04 (2.87) | -23.92 (9.22) | -39.39 (2.86)
  Week 228 (n=68, 5, 73) | -37.09 (2.96) | -17.60 (10.66) | -35.75 (2.89)
  Week 240 (n=65, 5, 70) | -38.91 (2.98) | -18.20 (8.36) | -37.43 (2.89)
  Week 252 (n=65, 5, 70) | -40.37 (2.92) | -7.60 (9.17) | -38.03 (2.95)
  Week 264 (n=59, 5, 64) | -37.32 (3.69) | -16.20 (9.01) | -35.67 (3.54)
  Week 276 (n=21, 1, 22) | -35.62 (6.09) | -10.00 (NA) — Standard error was not calculated due to one participant data available. | -34.45 (5.92)
  Week 288 (n=3, 0, 3) | -41.67 (7.31) | NA (NA) — Mean and standard error were not calculated because no data were available. | -41.67 (7.31)

8. Secondary Outcome: Change From Baseline in Physician Global Assessment of Arthritis
Description: Physician Global Assessment of Arthritis was measured on a 0 to 100 mm VAS, where 0 mm = very good and 100 mm = very bad. The baseline data of Study A3921039, A3921040 or A3921044 were used as baseline data for efficacy evaluations except for Modified Total Sharp Score (mTSS).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 2 (n= 378, 105, 483) | -42.80 (1.13) | -33.49 (2.01) | -40.78 (1.00)
  Week 4 (n=372, 105, 477) | -46.06 (1.08) | -34.91 (2.20) | -43.60 (0.99)
  Week 8 (n=371, 105, 476) | -47.34 (1.06) | -37.15 (2.00) | -45.09 (0.95)
  Week 12 (n=370, 105, 475) | -47.78 (1.09) | -36.56 (2.33) | -45.30 (1.00)
  Week 24 (n=357, 104, 461) | -48.29 (1.07) | -41.26 (2.01) | -46.70 (0.95)
  Week 36 (n=339, 102, 441) | -49.28 (1.09) | -41.92 (2.01) | -47.58 (0.97)
  Week 48 (n=331, 102, 433) | -49.96 (1.13) | -45.28 (2.08) | -48.86 (1.00)
  Week 60 (n=323, 102, 425) | -49.89 (1.14) | -47.01 (2.05) | -49.20 (1.00)
  Week 72 (n=315, 99, 414) | -50.03 (1.14) | -45.70 (1.95) | -48.99 (0.99)
  Week 84 (n=309, 92, 401) | -50.61 (1.16) | -46.89 (2.17) | -49.75 (1.02)
  Week 96 (n=281, 87, 368) | -49.99 (1.28) | -48.16 (2.23) | -49.55 (1.11)
  Week 108 (n=259, 83, 342) | -49.62 (1.33) | -47.99 (2.56) | -49.22 (1.18)
  Week 120 (n=242, 80, 322) | -49.42 (1.47) | -47.76 (2.39) | -49.01 (1.26)
  Week 132 (n=231, 78, 309) | -49.99 (1.41) | -50.19 (2.33) | -50.04 (1.20)
  Week 144 (n=224, 76, 300) | -50.80 (1.46) | -49.55 (2.44) | -50.49 (1.25)
  Week 156 (n=219, 72, 291) | -50.68 (1.39) | -49.78 (2.58) | -50.46 (1.23)
  Week 168 (n=213, 70, 283) | -51.52 (1.45) | -46.33 (2.60) | -50.23 (1.27)
  Week 180 (n=180, 57, 237) | -52.20 (1.51) | -50.33 (2.84) | -51.75 (1.33)
  Week 192 (n=138, 42, 180) | -51.41 (1.72) | -50.43 (2.98) | -51.18 (1.49)
  Week 204 (n=109, 30, 139) | -51.10 (1.73) | -50.97 (4.12) | -51.07 (1.61)
  Week 216 (n=76, 13, 89) | -50.91 (2.01) | -42.77 (6.37) | -49.72 (1.96)
  Week 228 (n=67, 5, 72) | -49.57 (2.37) | -33.60 (8.88) | -48.46 (2.33)
  Week 240 (n=65, 5, 70) | -49.94 (2.25) | -34.40 (10.30) | -48.83 (2.25)
  Week 252 (n=65, 5, 70) | -51.78 (2.17) | -31.60 (7.92) | -50.34 (2.17)
  Week 264 (n=58, 5, 63) | -52.62 (2.36) | -33.80 (9.49) | -51.13 (2.36)
  Week 276 (n=21, 1, 22) | -53.05 (3.92) | -7.00 (NA) — Standard error was not calculated due to one participant data available. | -50.95 (4.29)
  Week 288 (n=3, 0, 3) | -37.67 (1.33) | NA (NA) — Mean and standard error were not calculated because no data were available. | -37.67 (1.33)

9. Secondary Outcome: Change From Baseline in Patient Assessment of Arthritis Pain
Description: Participants rated the severity of arthritis pain on a 0 to 100 millimeter (mm) visual analogue scale (VAS), where 0 mm = no pain and 100 mm = most severe pain. The baseline data of Study A3921039, A3921040 or A3921044 were used as baseline data for efficacy evaluations except for Modified Total Sharp Score (mTSS).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 2 (n= 378, 105, 483) | -34.23 (1.40) | -27.98 (2.39) | -32.87 (1.22)
  Week 4 (n=372, 105, 477) | -37.32 (1.38) | -27.70 (2.61) | -35.20 (1.23)
  Week 8 (n=371, 105, 476) | -39.54 (1.34) | -30.69 (2.32) | -37.59 (1.17)
  Week 12 (n=370, 105, 475) | -39.34 (1.36) | -29.03 (2.25) | -37.06 (1.18)
  Week 24 (n=357, 104, 461) | -40.70 (1.42) | -33.60 (2.50) | -39.10 (1.24)
  Week 36 (n=339, 102, 441) | -41.70 (1.45) | -32.71 (2.56) | -39.62 (1.27)
  Week 48 (n=331, 102, 433) | -41.98 (1.41) | -34.39 (2.52) | -40.19 (1.24)
  Week 60 (n=323, 102, 425) | -42.37 (1.44) | -36.65 (2.36) | -41.00 (1.24)
  Week 72 (n=315, 99, 414) | -41.84 (1.51) | -37.41 (2.28) | -40.79 (1.28)
  Week 84 (n=309, 92, 401) | -42.49 (1.53) | -37.65 (2.55) | -41.38 (1.32)
  Week 96 (n=281, 87, 368) | -42.21 (1.63) | -38.21 (2.87) | -41.27 (1.42)
  Week 108 (n=259, 84, 343) | -42.61 (1.68) | -37.99 (2.87) | -41.48 (1.45)
  Week 120 (n=242, 80, 322) | -42.44 (1.74) | -37.45 (2.92) | -41.20 (1.50)
  Week 132 (n=232, 79, 311) | -42.52 (1.78) | -37.86 (3.04) | -41.33 (1.54)
  Week 144 (n=224, 76, 300) | -42.05 (1.81) | -37.07 (3.09) | -40.79 (1.56)
  Week 156 (n=219, 72, 291) | -43.77 (1.75) | -36.39 (2.89) | -41.94 (1.51)
  Week 168 (n=213, 70, 283) | -43.87 (1.73) | -37.96 (3.24) | -42.41 (1.54)
  Week 180 (n=180, 57, 237) | -43.85 (1.92) | -40.21 (3.51) | -42.97 (1.68)
  Week 192 (n=138, 42, 180) | -42.64 (2.22) | -36.67 (3.93) | -41.24 (1.94)
  Week 204 (n=109, 30, 139) | -41.11 (2.59) | -38.70 (5.25) | -40.59 (2.32)
  Week 216 (n=76, 13, 89) | -41.61 (2.90) | -30.38 (9.30) | -39.97 (2.84)
  Week 228 (n=68, 5, 73) | -37.19 (2.96) | -28.40 (12.48) | -36.59 (2.87)
  Week 240 (n=65, 5, 70) | -36.72 (3.08) | -21.20 (7.85) | -35.61 (2.94)
  Week 252 (n=65, 5, 70) | -38.54 (3.19) | -21.20 (10.56) | -37.30 (3.08)
  Week 264 (n=59, 5, 64) | -36.80 (3.72) | -16.60 (11.91) | -35.22 (3.60)
  Week 276 (n=21, 1, 22) | -40.19 (5.00) | -44.00 (NA) — Standard error was not calculated due to one participant data available. | -40.36 (4.77)
  Week 288 (n=3, 0, 3) | -34.67 (9.82) | NA (NA) — Mean and standard error were not calculated because no data were available. | -34.67 (9.82)

10. Secondary Outcome: Change From Baseline in Tender/Painful Joint Counts
Description: This was carried out on 68 joints. Each joint's response to pressure/motion was assessed using the following scale: Present/Absent/Not Done/Not Applicable (to be used for artificial joints). The baseline data of Study A3921039, A3921040 or A3921044 were used as baseline data for efficacy evaluations except for Modified Total Sharp Score (mTSS).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Tender/painful joints
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Tender/painful joints
  Week 2 (n=378, 105, 483) | -11.88 (0.48) | -10.17 (0.95) | -11.51 (0.43)
  Week 4 (n=373, 105, 478) | -12.13 (0.51) | -10.46 (0.90) | -11.77 (0.45)
  Week 8 (n=371, 105, 476) | -13.06 (0.47) | -10.75 (0.96) | -12.55 (0.43)
  Week 12 (n=370, 105, 475) | -13.41 (0.47) | -10.74 (0.97) | -12.82 (0.43)
  Week 24 (n=357, 104, 461) | -14.02 (0.50) | -12.62 (0.89) | -13.70 (0.44)
  Week 36 (n=339, 102, 441) | -14.32 (0.53) | -13.05 (0.94) | -14.03 (0.46)
  Week 48 (n=331, 102, 433) | -14.23 (0.53) | -13.43 (0.99) | -14.04 (0.47)
  Week 60 (n=323, 102, 425) | -14.23 (0.55) | -13.67 (0.94) | -14.09 (0.48)
  Week 72 (n=315, 99, 414) | -14.45 (0.56) | -14.00 (0.96) | -14.34 (0.48)
  Week 84 (n=309, 92, 401) | -14.39 (0.56) | -14.04 (1.11) | -14.31 (0.50)
  Week 96 (n=281, 87, 368) | -14.44 (0.60) | -13.92 (1.03) | -14.32 (0.52)
  Week 108 (n=259, 83, 342) | -14.46 (0.61) | -13.66 (1.14) | -14.26 (0.54)
  Week 120 (n=242, 80, 322) | -14.67 (0.65) | -13.69 (1.07) | -14.42 (0.55)
  Week 132 (n=232, 79, 311) | -14.01 (0.73) | -13.30 (1.33) | -13.83 (0.64)
  Week 144 (n=224, 76, 300) | -14.45 (0.68) | -13.83 (1.18) | -14.29 (0.59)
  Week 156 (n=219, 72, 291) | -14.24 (0.70) | -14.15 (1.20) | -14.22 (0.61)
  Week 168 (n=213, 70, 283) | -14.41 (0.73) | -14.06 (1.25) | -14.33 (0.63)
  Week 180 (n=180, 57, 237) | -14.78 (0.79) | -15.18 (1.46) | -14.87 (0.70)
  Week 192 (n=138, 42, 180) | -15.01 (0.87) | -14.57 (1.42) | -14.91 (0.74)
  Week 204 (n=109, 30, 139) | -14.79 (0.94) | -15.67 (1.93) | -14.98 (0.84)
  Week 216 (n=76, 13, 89) | -14.42 (1.04) | -11.38 (2.64) | -13.98 (0.97)
  Week 228 (n=68, 5, 73) | -13.78 (1.56) | -11.60 (5.46) | -13.63 (1.49)
  Week 240 (n=65, 5, 70) | -15.11 (1.15) | -10.80 (4.92) | -14.80 (1.12)
  Week 252 (n=65, 5, 70) | -15.34 (1.17) | -9.60 (4.55) | -14.93 (1.14)
  Week 264 (n=59, 5, 64) | -15.54 (1.27) | -9.80 (3.95) | -15.09 (1.22)
  Week 276 (n=22, 1, 23) | -17.55 (2.55) | -4.00 (NA) — Standard error was not calculated due to one participant data available. | -16.96 (2.51)
  Week 288 (n=3, 0, 3) | -8.67 (1.20) | NA (NA) — Mean and standard error were not calculated because no data were available. | -8.67 (1.20)

11. Secondary Outcome: Change From Baseline in Swollen Joint Counts
Description: Sixty-six (66) joints, the same as those assessed for tenderness/pain except for the right and left hip joints, were assessed for swelling by palpation using the following scale: Present/Absent/Not Done/Not Applicable (to be used for artificial joints). The baseline data of Study A3921039, A3921040 or A3921044 were used as baseline data for efficacy evaluations except for Modified Total Sharp Score (mTSS).
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Swollen joints
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Swollen joints
  Week 2 (n=378, 105, 483) | -9.67 (0.38) | -8.69 (0.74) | -9.46 (0.34)
  Week 4 (n=373, 105, 478) | -10.12 (0.42) | -8.54 (0.75) | -9.78 (0.37)
  Week 8 (n=371, 105, 476) | -10.90 (0.39) | -9.31 (0.73) | -10.55 (0.35)
  Week 12 (n=370, 105, 475) | -11.18 (0.40) | -9.21 (0.67) | -10.74 (0.35)
  Week 24 (n=357, 104, 461) | -11.33 (0.40) | -10.46 (0.72) | -11.13 (0.35)
  Week 36 (n=339, 102, 441) | -11.62 (0.43) | -10.75 (0.73) | -11.41 (0.37)
  Week 48 (n=331, 102, 433) | -11.76 (0.44) | -11.11 (0.74) | -11.61 (0.38)
  Week 60 (n=323, 102, 425) | -11.83 (0.44) | -10.97 (0.76) | -11.62 (0.38)
  Week 72 (n=315, 99, 414) | -12.00 (0.46) | -11.38 (0.80) | -11.85 (0.40)
  Week 84 (n=309, 92, 401) | -12.08 (0.47) | -11.72 (0.88) | -12.00 (0.41)
  Week 96 (n=281, 87, 368) | -11.97 (0.50) | -11.54 (0.84) | -11.87 (0.43)
  Week 108 (n=259, 83, 342) | -11.94 (0.52) | -11.60 (0.91) | -11.86 (0.45)
  Week 120 (n=242, 80, 322) | -12.09 (0.56) | -11.24 (0.87) | -11.88 (0.47)
  Week 132 (n=232, 79, 311) | -11.69 (0.64) | -11.15 (1.16) | -11.55 (0.56)
  Week 144 (n=224, 76, 300) | -11.90 (0.61) | -11.74 (0.94) | -11.86 (0.51)
  Week 156 (n=219, 72, 291) | -12.07 (0.61) | -11.86 (1.04) | -12.02 (0.52)
  Week 168 (n=213, 70, 283) | -12.17 (0.62) | -11.67 (1.05) | -12.05 (0.54)
  Week 180 (n=180, 57, 237) | -12.43 (0.70) | -12.26 (1.24) | -12.39 (0.61)
  Week 192 (n=138, 42, 180) | -12.36 (0.79) | -12.48 (1.47) | -12.38 (0.69)
  Week 204 (n=109, 30, 139) | -12.35 (0.82) | 12.50 (1.89) | 12.38 (0.76)
  Week 216 (n=76, 13, 89) | -12.34 (0.99) | -9.00 (2.35) | -11.85 (0.91)
  Week 228 (n=68, 5, 73) | -11.74 (1.47) | -11.00 (5.09) | -11.68 (1.41)
  Week 240 (n=65, 5, 70) | -13.09 (1.12) | -11.40 (5.48) | -12.97 (1.10)
  Week 252 (n=65, 5, 70) | -13.20 (1.15) | -10.60 (4.70) | -13.01 (1.11)
  Week 264 (n=59, 5, 64) | -13.58 (1.24) | -10.00 (4.11) | -13.30 (1.19)
  Week 276 (n=22, 1, 23) | -15.32 (2.53) | -6.00 (NA) — Standard error was not calculated due to one participant data available. | -14.91 (2.46)
  Week 288 (n=3, 0, 3) | -8.33 (0.88) | NA (NA) — Mean and standard error were not calculated because no data were available. | -8.33 (0.88)

12. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Domain Score_Physical Functioning
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning) and is reported as 2 summary scores; physical component score and mental component score. Total score range for the summary scores = 0-100, where higher score represents higher level of functioning. The baseline data of Study A3921039, A3921040 or A3921044 were used as baseline data for efficacy evaluations except for Modified Total Sharp Score (mTSS).
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 12 (n=370, 105, 475) | 7.87 (0.45) | 5.94 (0.76) | 7.45 (0.39)
  Week 24 (n=357, 104, 461) | 8.67 (0.46) | 6.12 (1.01) | 8.10 (0.42)
  Week 48 (n=331, 102, 433) | 9.06 (0.48) | 6.84 (1.05) | 8.54 (0.45)
  Week 72 (n=315, 99, 414) | 9.10 (0.51) | 7.61 (0.93) | 8.74 (0.45)
  Week 96 (n=281, 87, 368) | 9.11 (0.55) | 8.26 (0.88) | 8.91 (0.47)
  Week 120 (n=242, 80, 322) | 9.12 (0.57) | 8.34 (1.09) | 8.92 (0.51)
  Week 144 (n=224, 76, 300) | 8.85 (0.66) | 7.57 (1.18) | 8.53 (0.57)
  Week 168 (n=213, 70, 283) | 9.01 (0.68) | 7.16 (1.36) | 8.55 (0.61)
  Week 192 (n=138, 42, 180) | 9.43 (0.78) | 8.09 (1.25) | 9.12 (0.66)
  Week 216 (n=76, 13, 89) | 8.78 (0.98) | 5.04 (2.27) | 8.23 (0.91)
  Week 240 (n=65, 5, 70) | 8.91 (1.00) | 3.27 (1.90) | 8.51 (0.95)
  Week 264 (n=59, 5, 64) | 8.85 (1.08) | 1.64 (1.98) | 8.28 (1.03)
  Week 288 (n=3, 0, 3) | 10.23 (1.18) | NA (NA) — Mean and standard error were not calculated because no data were available. | 10.23 (1.18)

13. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Domain Score_Role Physical
Description: as for outcome 12
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 12 (n=370, 105, 475) | 7.31 (0.57) | 5.48 (1.00) | 6.90 (0.50)
  Week 24 (n=357, 104, 461) | 8.21 (0.59) | 6.29 (1.06) | 7.77 (0.51)
  Week 48 (n=331, 102, 433) | 8.38 (0.64) | 7.77 (0.92) | 8.23 (0.53)
  Week 72 (n=315, 99, 414) | 7.23 (0.67) | 7.47 (1.08) | 7.29 (0.57)
  Week 96 (n=281, 87, 368) | 7.24 (0.70) | 8.15 (1.16) | 7.46 (0.60)
  Week 120 (n=242, 80, 322) | 7.69 (0.75) | 6.77 (1.10) | 7.46 (0.63)
  Week 144 (n=224, 76, 300) | 7.21 (0.80) | 6.56 (1.23) | 7.05 (0.67)
  Week 168 (n=213, 70, 283) | 7.38 (0.77) | 5.42 (1.41) | 6.90 (0.68)
  Week 192 (n=138, 42, 180) | 6.59 (1.01) | 6.70 (1.57) | 6.61 (0.86)
  Week 216 (n=76, 13, 89) | 6.53 (1.37) | 4.59 (2.53) | 6.25 (1.22)
  Week 240 (n=65, 5, 70) | 6.13 (1.56) | -0.48 (2.86) | 5.66 (1.48)
  Week 264 (n=59, 5, 64) | 6.15 (1.58) | 0.95 (2.68) | 5.74 (1.48)
  Week 288 (n=3, 0, 3) | 22.27 (5.22) | NA (NA) — Mean and standard error were not calculated because no data were available. | 22.27 (5.22)

14. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Domain Score_Bodily Pain
Description: as for outcome 12
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 12 (n=370, 105, 475) | 11.40 (0.48) | 8.13 (0.77) | 10.40 (0.41)
  Week 24 (n=357, 104, 461) | 11.87 (0.50) | 9.63 (0.79) | 11.36 (0.43)
  Week 48 (n=331, 102, 433) | 12.19 (0.53) | 10.65 (0.75) | 11.83 (0.44)
  Week 72 (n=315, 99, 414) | 11.96 (0.56) | 9.92 (0.81) | 11.47 (0.47)
  Week 96 (n=281, 87, 368) | 11.35 (0.59) | 11.60 (1.04) | 11.41 (0.51)
  Week 120 (n=242, 80, 322) | 11.98 (0.62) | 10.42 (1.08) | 11.60 (0.54)
  Week 144 (n=224, 76, 300) | 11.51 (0.68) | 11.15 (1.04) | 11.42 (0.57)
  Week 168 (n=213, 70, 283) | 11.82 (0.65) | 11.07 (1.11) | 11.63 (0.56)
  Week 192 (n=138, 42, 180) | 11.19 (0.85) | 11.43 (1.57) | 11.25 (0.75)
  Week 216 (n=76, 13, 89) | 12.43 (1.03) | 8.52 (2.37) | 11.86 (0.95)
  Week 240 (n=65, 5, 70) | 11.34 (1.04) | 5.25 (2.63) | 10.90 (0.99)
  Week 264 (n=59, 5, 64) | 11.27 (1.28) | 4.50 (2.87) | 10.74 (1.22)
  Week 288 (n=3, 0, 3) | 7.08 (5.60) | NA (NA) — Mean and standard error were not calculated because no data were available. | 7.08 (5.60)

15. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Domain Score_General Health
Description: as for outcome 12
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 12 (n=370, 105, 475) | 6.07 (0.38) | 4.24 (0.70) | 5.67 (0.34)
  Week 24 (n=357, 104, 461) | 6.38 (0.39) | 5.00 (0.58) | 6.07 (0.33)
  Week 48 (n=331, 102, 433) | 6.40 (0.40) | 5.20 (0.67) | 6.12 (0.34)
  Week 72 (n=315, 99, 414) | 6.29 (0.42) | 5.35 (0.63) | 6.06 (0.35)
  Week 96 (n=281, 87, 368) | 6.00 (0.45) | 4.82 (0.73) | 5.72 (0.38)
  Week 120 (n=242, 80, 322) | 5.86 (0.49) | 5.36 (0.82) | 5.74 (0.42)
  Week 144 (n=224, 76, 300) | 5.37 (0.54) | 4.38 (0.94) | 5.12 (0.47)
  Week 168 (n=213, 70, 283) | 5.82 (0.53) | 3.93 (0.87) | 5.35 (0.46)
  Week 192 (n=138, 42, 180) | 4.72 (0.61) | 4.10 (1.05) | 4.57 (0.53)
  Week 216 (n=76, 13, 89) | 3.73 (0.87) | 1.59 (1.31) | 3.42 (0.77)
  Week 240 (n=65, 5, 70) | 4.39 (0.96) | -1.50 (1.90) | 3.97 (0.92)
  Week 264 (n=59, 5, 64) | 4.12 (1.01) | -1.03 (2.17) | 3.72 (0.96)
  Week 288 (n=3, 0, 3) | -0.94 (4.23) | NA (NA) — Mean and standard error were not calculated because no data were available. | -0.94 (4.23)

16. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Domain Score_Vitality
Description: as for outcome 12
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 12 (n=370, 105, 475) | 7.37 (0.59) | 6.61 (0.90) | 7.20 (0.50)
  Week 24 (n=357, 104, 461) | 7.24 (0.58) | 6.25 (0.97) | 7.02 (0.50)
  Week 48 (n=331, 102, 433) | 6.83 (0.58) | 7.22 (0.89) | 6.92 (0.49)
  Week 72 (n=315, 99, 414) | 7.02 (0.61) | 6.44 (0.98) | 6.88 (0.52)
  Week 96 (n=281, 87, 368) | 6.78 (0.61) | 6.19 (1.11) | 6.64 (0.54)
  Week 120 (n=242, 80, 322) | 6.49 (0.70) | 6.96 (1.26) | 6.61 (0.61)
  Week 144 (n=224, 76, 300) | 6.27 (0.75) | 5.51 (1.15) | 6.08 (0.63)
  Week 168 (n=213, 70, 283) | 6.58 (0.72) | 4.75 (1.27) | 6.12 (0.63)
  Week 192 (n=138, 42, 180) | 5.40 (0.92) | 5.70 (1.62) | 5.47 (0.80)
  Week 216 (n=76, 13, 89) | 5.04 (1.18) | 5.30 (2.47) | 5.08 (1.07)
  Week 240 (n=65, 5, 70) | 5.11 (1.21) | -0.60 (3.05) | 4.70 (1.15)
  Week 264 (n=59, 5, 64) | 4.72 (1.17) | -1.80 (3.36) | 4.21 (1.13)
  Week 288 (n=3, 0, 3) | 14.97 (8.64) | NA (NA) — Mean and standard error were not calculated because no data were available. | 14.97 (8.64)

17. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Domain Score_Social Functioning
Description: as for outcome 12
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 12 (n=370, 105, 475) | 4.99 (0.60) | 5.17 (1.09) | 5.03 (0.52)
  Week 24 (n=357, 104, 461) | 5.57 (0.62) | 4.96 (1.25) | 5.44 (0.56)
  Week 48 (n=331, 102, 433) | 5.28 (0.64) | 5.27 (1.14) | 5.28 (0.55)
  Week 72 (n=315, 99, 414) | 4.81 (0.64) | 4.78 (1.31) | 4.81 (0.58)
  Week 96 (n=281, 87, 368) | 4.88 (0.67) | 6.43 (1.19) | 5.25 (0.58)
  Week 120 (n=242, 80, 322) | 5.20 (0.76) | 5.98 (1.11) | 5.39 (0.63)
  Week 144 (n=224, 76, 300) | 5.23 (0.77) | 3.33 (1.39) | 4.75 (0.67)
  Week 168 (n=213, 70, 283) | 4.72 (0.79) | 3.84 (1.43) | 4.50 (0.69)
  Week 192 (n=138, 42, 180) | 4.56 (0.96) | 5.63 (1.36) | 4.81 (0.80)
  Week 216 (n=76, 13, 89) | 4.53 (1.23) | 3.31 (2.48) | 4.35 (1.10)
  Week 240 (n=65, 5, 70) | 4.88 (1.41) | 0.00 (0.00) | 4.53 (1.32)
  Week 264 (n=59, 5, 64) | 4.47 (1.45) | -2.15 (2.15) | 3.95 (1.37)
  Week 288 (n=3, 0, 3) | 14.34 (9.49) | NA (NA) — Mean and standard error were not calculated because no data were available. | 14.34 (9.49)

18. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Domain Score_Role Emotional
Description: as for outcome 12
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 12 (n=370, 105, 475) | 6.65 (0.65) | 4.98 (1.19) | 6.28 (0.57)
  Week 24 (n=357, 104, 461) | 6.88 (0.73) | 4.40 (1.41) | 6.32 (0.65)
  Week 48 (n=331, 102, 433) | 7.26 (0.75) | 5.49 (1.29) | 6.85 (0.65)
  Week 72 (n=315, 99, 414) | 6.02 (0.78) | 5.54 (1.28) | 5.91 (0.67)
  Week 96 (n=281, 87, 368) | 6.04 (0.79) | 5.96 (1.43) | 6.02 (0.69)
  Week 120 (n=242, 80, 322) | 5.68 (0.90) | 3.98 (1.40) | 5.26 (0.76)
  Week 144 (n=224, 76, 300) | 5.39 (0.96) | 3.74 (1.56) | 4.97 (0.82)
  Week 168 (n=213, 70, 283) | 5.90 (0.89) | 4.43 (1.49) | 5.54 (0.76)
  Week 192 (n=138, 42, 180) | 4.31 (1.23) | 4.42 (1.91) | 4.33 (1.04)
  Week 216 (n=76, 13, 89) | 4.33 (1.55) | 3.49 (2.76) | 4.21 (1.38)
  Week 240 (n=65, 5, 70) | 4.72 (1.66) | -0.76 (4.22) | 4.33 (1.58)
  Week 264 (n=59, 5, 64) | 5.07 (1.74) | -0.76 (4.22) | 4.61 (1.64)
  Week 288 (n=3, 0, 3) | 22.71 (5.78) | NA (NA) — Mean and standard error were not calculated because no data were available. | 22.71 (5.78)

19. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Domain Score_Mental Health
Description: as for outcome 12
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 12 (n=370, 105, 475) | 6.27 (0.63) | 5.38 (1.04) | 6.08 (0.54)
  Week 24 (n=357, 104, 461) | 6.22 (0.65) | 3.84 (1.17) | 5.69 (0.57)
  Week 48 (n=331, 102, 433) | 5.73 (0.64) | 5.35 (1.02) | 5.64 (0.54)
  Week 72 (n=315, 99, 414) | 4.77 (0.70) | 5.48 (1.04) | 4.94 (0.59)
  Week 96 (n=281, 87, 368) | 5.23 (0.68) | 5.89 (1.14) | 5.38 (0.59)
  Week 120 (n=242, 80, 322) | 5.56 (0.77) | 5.26 (1.31) | 5.49 (0.67)
  Week 144 (n=224, 76, 300) | 5.10 (0.84) | 4.37 (1.34) | 4.91 (0.71)
  Week 168 (n=213, 70, 283) | 5.12 (0.76) | 3.76 (1.29) | 4.79 (0.66)
  Week 192 (n=138, 42, 180) | 3.77 (0.93) | 5.21 (1.75) | 4.11 (0.82)
  Week 216 (n=76, 13, 89) | 2.66 (1.21) | 4.26 (3.04) | 2.89 (1.12)
  Week 240 (n=65, 5, 70) | 3.75 (1.20) | 3.32 (2.04) | 3.72 (1.12)
  Week 264 (n=59, 5, 64) | 4.18 (1.34) | 0.00 (1.75) | 3.85 (1.25)
  Week 288 (n=3, 0, 3) | 14.78 (7.56) | NA (NA) — Mean and standard error were not calculated because no data were available. | 14.78 (7.56)

20. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Component Score_Physical
Description: as for outcome 12
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 12 (n=370, 105, 475) | 8.44 (0.39) | 6.09 (0.68) | 7.92 (0.34)
  Week 24 (n=357, 104, 461) | 9.39 (0.38) | 7.56 (0.70) | 8.98 (0.34)
  Week 48 (n=331, 102, 433) | 9.75 (0.43) | 8.24 (0.72) | 9.39 (0.37)
  Week 72 (n=315, 99, 414) | 9.72 (0.43) | 8.21 (0.76) | 9.36 (0.37)
  Week 96 (n=281, 87, 368) | 9.35 (0.48) | 8.93 (0.77) | 9.25 (0.41)
  Week 120 (n=242, 80, 322) | 9.66 (0.49) | 8.79 (0.92) | 9.45 (0.43)
  Week 144 (n=224, 76, 300) | 9.26 (0.54) | 8.60 (0.92) | 9.09 (0.47)
  Week 168 (n=213, 70, 283) | 9.51 (0.54) | 7.86 (1.03) | 9.10 (0.48)
  Week 192 (n=138, 42, 180) | 9.51 (0.65) | 8.56 (1.18) | 9.29 (0.57)
  Week 216 (n=76, 13, 89) | 9.59 (0.88) | 5.37 (1.93) | 8.97 (0.82)
  Week 240 (n=65, 5, 70) | 9.00 (0.93) | 1.91 (2.87) | 8.49 (0.91)
  Week 264 (n=59, 5, 64) | 8.72 (1.03) | 2.31 (2.27) | 8.22 (0.99)
  Week 288 (n=3, 0, 3) | 6.87 (1.88) | NA (NA) — Mean and standard error were not calculated because no data were available. | 6.87 (1.88)

21. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Component Score_Mental
Description: as for outcome 12
Time Frame: Baseline, Weeks 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Units on a scale
  Week 12 (n=370, 105, 475) | 5.13 (0.63) | 4.82 (1.01) | 5.06 (0.54)
  Week 24 (n=357, 104, 461) | 4.95 (0.67) | 3.38 (1.26) | 4.60 (0.59)
  Week 48 (n=331, 102, 433) | 4.56 (0.66) | 4.45 (1.06) | 4.54 (0.56)
  Week 72 (n=315, 99, 414) | 3.63 (0.69) | 4.15 (1.14) | 3.75 (0.59)
  Week 96 (n=281, 87, 368) | 3.88 (0.68) | 4.53 (1.25) | 4.03 (0.60)
  Week 120 (n=242, 80, 322) | 3.79 (0.80) | 3.68 (1.37) | 3.76 (0.69)
  Week 144 (n=224, 76, 300) | 3.57 (0.84) | 2.24 (1.40) | 3.23 (0.72)
  Week 168 (n=213, 70, 283) | 3.64 (0.80) | 2.45 (1.41) | 3.35 (0.70)
  Week 192 (n=138, 42, 180) | 2.05 (0.99) | 3.44 (1.80) | 2.38 (0.86)
  Week 216 (n=76, 13, 89) | 1.49 (1.29) | 3.14 (3.04) | 1.73 (1.18)
  Week 240 (n=65, 5, 70) | 2.41 (1.27) | -0.04 (1.81) | 2.23 (1.19)
  Week 264 (n=59, 5, 64) | 2.59 (1.42) | -2.25 (1.41) | 2.21 (1.32)
  Week 288 (n=3, 0, 3) | 18.64 (4.01) | NA (NA) — Mean and standard error were not calculated because no data were available. | 18.64 (4.01)

22. Secondary Outcome: Change From Month 24 in Study A3921044 in Modified Total Sharp Score (mTSS)
Description: mTSS = sum of erosion and Joint Space Narrowing (JSN) scores for 44 joints (16 per hand and 6 per foot). mTSS scores range from 0 (normal) to 448 (worst possible total score). Change: scores at observation minus score at baseline. An increase in mTSS from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented potential improvement. Month 24 (the final visit) in Study A3921044 was taken as the first visit in current study.
Time Frame: First visit in the study (Month 24 in Study A3921044), Weeks 24, 48, and 96
Population: Participants who had completed Study A3921044 among all participants who received at least 1 dose of study medication in current study. No imputation was used (observed data).
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 75 | 7 | 82
Units on a scale
  Week 24 (n=69, 7, 76) | 0.17 (0.09) | 0.50 (0.22) | 0.20 (0.08)
  Week 48 (n=64, 7, 71) | 0.27 (0.17) | 1.75 (1.16) | 0.41 (0.19)
  Week 96 (n=39, 1, 40) | 0.40 (0.21) | 1.00 (NA) — Standard error was not calculated because there was one participant data. | 0.42 (0.20)

23. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to the last participants visit in the study. The baseline data of Study A3921039, A3921040 or A3921044 were used as baseline data for safety evaluation.
Time Frame: Baseline up to Week 288
Population: Safety analysis set: all participants who received at least 1 dose of study medication in current study.
Measure: Number; unit: Particiants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 381 | 105 | 486
Particiants
  Number of participants with AEs (including SAEs) | 371 | 105 | 476
  Number of participants with SAEs | 111 | 28 | 139

ADVERSE EVENTS:
Time Frame: Safety observations up to Week 288
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Serious Adverse Events (participants affected / at risk) | 111/381 | 28/105 | 139/486
Other Adverse Events (participants affected / at risk) | 345/381 | 101/105 | 446/486
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg BID (N=381) | CP-690,550 10 mg BID (N=105) | Total (N=486)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Prinzmetal angina (Cardiac disorders) | 1 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 1
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0 | 1
Cataract (Eye disorders) | 2 | 1 | 3
Dacryostenosis acquired (Eye disorders) | 1 | 0 | 1
Retinal artery occlusion (Eye disorders) | 0 | 1 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Large intestine polyp (Gastrointestinal disorders) | 3 | 0 | 3
Radicular cyst (Gastrointestinal disorders) | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 1
Device material issue (General disorders) | 1 | 0 | 1
Submandibular mass (General disorders) | 0 | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 3 | 1 | 4
Chronic sinusitis (Infections and infestations) | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 1
Enteritis infectious (Infections and infestations) | 1 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 1
Enterocolitis viral (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 1 | 3
Herpes zoster (Infections and infestations) | 11 | 2 | 13
Herpes zoster disseminated (Infections and infestations) | 0 | 1 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 0 | 2
Pneumonia (Infections and infestations) | 6 | 1 | 7
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 2 | 0 | 2
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 3 | 2 | 5
Sepsis (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 0 | 2
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 9 | 0 | 9
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Computerised tomogram thorax abnormal (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint destruction (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Periostitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 3
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Paget's disease of nipple (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 1
Cerebral thrombosis (Nervous system disorders) | 1 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 1
Cubital tunnel syndrome (Nervous system disorders) | 1 | 0 | 1
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1
Spondylitic myelopathy (Nervous system disorders) | 1 | 0 | 1
Temporal lobe epilepsy (Nervous system disorders) | 1 | 0 | 1
Transient global amnesia (Nervous system disorders) | 1 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 1 | 2
Glomerulonephritis membranous (Renal and urinary disorders) | 1 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg BID (N=381) | CP-690,550 10 mg BID (N=105) | Total (N=486)
Anaemia (Blood and lymphatic system disorders) | 14 | 11 | 25
Conjunctivitis (Eye disorders) | 17 | 6 | 23
Abdominal pain upper (Gastrointestinal disorders) | 13 | 6 | 19
Constipation (Gastrointestinal disorders) | 34 | 9 | 43
Dental caries (Gastrointestinal disorders) | 39 | 15 | 54
Diarrhoea (Gastrointestinal disorders) | 28 | 5 | 33
Gastritis (Gastrointestinal disorders) | 22 | 4 | 26
Stomatitis (Gastrointestinal disorders) | 25 | 7 | 32
Pyrexia (General disorders) | 15 | 9 | 24
Bronchitis (Infections and infestations) | 45 | 5 | 50
Cystitis (Infections and infestations) | 39 | 7 | 46
Gastroenteritis (Infections and infestations) | 34 | 11 | 45
Gingivitis (Infections and infestations) | 10 | 7 | 17
Herpes zoster (Infections and infestations) | 59 | 22 | 81
Influenza (Infections and infestations) | 37 | 11 | 48
Nasopharyngitis (Infections and infestations) | 221 | 72 | 293
Oral herpes (Infections and infestations) | 26 | 7 | 33
Periodontitis (Infections and infestations) | 20 | 3 | 23
Pharyngitis (Infections and infestations) | 36 | 10 | 46
Tinea pedis (Infections and infestations) | 31 | 3 | 34
Upper respiratory tract infection (Infections and infestations) | 40 | 8 | 48
Contusion (Injury, poisoning and procedural complications) | 36 | 12 | 48
Fall (Injury, poisoning and procedural complications) | 51 | 20 | 71
Ligament sprain (Injury, poisoning and procedural complications) | 11 | 9 | 20
Road traffic accident (Injury, poisoning and procedural complications) | 9 | 8 | 17
Alanine aminotransferase increased (Investigations) | 25 | 1 | 26
Aspartate aminotransferase increased (Investigations) | 22 | 1 | 23
Blood cholesterol increased (Investigations) | 9 | 6 | 15
Low density lipoprotein increased (Investigations) | 17 | 6 | 23
Lymphocyte count decreased (Investigations) | 29 | 9 | 38
White blood cell count decreased (Investigations) | 17 | 10 | 27
Hypercholesterolaemia (Metabolism and nutrition disorders) | 13 | 6 | 19
Hyperlipidaemia (Metabolism and nutrition disorders) | 36 | 20 | 56
Back pain (Musculoskeletal and connective tissue disorders) | 43 | 3 | 46
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 6 | 7 | 13
Headache (Nervous system disorders) | 38 | 10 | 48
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 9 | 33
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 4 | 23
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 25 | 9 | 34
Eczema (Skin and subcutaneous tissue disorders) | 25 | 2 | 27
Rash (Skin and subcutaneous tissue disorders) | 17 | 6 | 23
Hypertension (Vascular disorders) | 40 | 15 | 55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.